CLINICAL TRIAL: NCT03710928
Title: Type 1 Diabetes Management Using a Very Low Carbohydrate Versus Standard Diet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Belinda Lennerz, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00030039
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Type1diabetes
Keywords: very low carbohydrate diet; nutrition; ketogenic diet; ketosis; nutritional ketosis; metabolism; metabolic health
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: randomized controlled trial, 12-week feeding study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- very low carbohydrate diet (Experimental): Dietary Intervention, food delivery
  Interventions: Other: very low carbohydrate diet
- standard diet (Active Comparator): Dietary Intervention, food delivery
  Interventions: Other: standard carbohydrate diet

INTERVENTIONS:
Other: very low carbohydrate diet — All meals will be delivered and participants will consume study foods exclusively. Participants will receive a fiber supplement as needed with each meal to support digestive health, and a daily multi-vitamin, magnesium and omega-three supplement to ascertain micronutrient sufficiency. Participants will be weighed at each study visit and the diet plan will be adjusted for satiety and weight-maintenance.
  The diet composition will be as follows: 5% carbohydrate, 70% fat, 20% protein.
  Arms: very low carbohydrate diet
Other: standard carbohydrate diet — All meals will be delivered and participants will consume study foods exclusively. Participants will receive a daily multi-vitamin and omega-3 supplement to ascertain micronutrient sufficiency. Participants will be weighed at each study visit and the diet plan will be adjusted for satiety and weight-maintenance.
  The diet composition will be as follows: 50% carbohydrate, 30% fat, 20% protein.
  Arms: standard diet

SUMMARY:
Despite major technological advances, management of type one diabetes mellitus (T1D) remains suboptimal, putting millions of people at risk for immediate and long-term complications. After meals, a mismatch between carbohydrate absorption rate and insulin action typically leads to alternating periods of hyper- and hypoglycemia. A conceptually promising approach to control both problems is dietary carbohydrate restriction to reduce postprandial blood glucose changes and insulin needs. In a prior survey study, the investigators documented exceptional glycemic control (HbA1c 5.67%) and low acute complication rates among 316 children and adults with T1D consuming a very-low-carbohydrate diet.

To test the feasibility of this approach, the investigators will conduct a randomized-controlled feeding study involving 32 adults and adolescents with T1D. Participants will be randomized to receive a very low carbohydrate vs. standard carbohydrate diet. Participants will be in the study for 12 weeks and receive all their meals by meal delivery.They will share continuous glucose monitoring data with the study team and be in close communication to adjust insulin doses as needed. All participants will have a screening visit, an individual or group education session, and 3 study visits to evaluate diabetes control and metabolic health. Some of these visits will have a fasting blood draw. Two of the visits will also comprise additional metabolic studies to assess glucagon response and brain function during hypoglycemia by magnetic resonance imaging (MRI). Participants will have IV catheters placed and receive IV insulin to drop blood glucose levels to 50 mg/dl for up to 30 minutes. The primary outcome will be HbA1c change from baseline. Secondary outcomes include detailed measures of glycemic variability, metabolic health, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with T1D for at least 1 year
* Age 18 to 40 years
* Tanner stage ≥ IV
* BMI 18.5-35 kg/m2
* Stable glycemic control (HbA1c 6.5-9%)
* Use of a continuous glucose monitor (CGM)
* Use of an insulin pump
* Attendance of at least 1 diabetes care visit over the past 12 months (including virtual)

Exclusion Criteria:

* Ketoacidosis or severe hypoglycemia with seizure or coma in the past 6 months
* Dietary restrictions or intolerances that are incompatible with the planned food deliveries, e.g. celiac disease, gastroparesis, certain food allergies
* Following a weight-loss or otherwise restrictive diet
* Vigorous exercise >2 hours on >3 days a week
* History of an eating disorder or at risk for eating disorder, assessed by the Eating Disorders Diagnostic Scale (EDDS)
* Major medical illness or use of medications other than insulin and metformin that could interfere with metabolic or glycemic variables
* Significant psychiatric illness
* Smoking, use of recreational drugs, or excessive alcohol consumption
* Pregnancy or breastfeeding
* Anemia
* For participants who undergo MRI:

  1. Standard MRI exclusion criteria
  2. Irregular menses
  3. Use of psychotropic medication other than SSRIs or other mild antidepressant or anxiety medications (unless these medications are safe to be held for several days to allow for the acquisition of MRI data)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C change | 12 weeks - baseline
  HbA1C change from baseline at 12 weeks will be compared between the 2 interventions

SECONDARY OUTCOMES:
total daily insulin dose | week 0 and 12
  average daily insulin dose over 1 week will be calculated
percent time spent in the glycemic target range of 70-140 mg/dl | week 0 and 12
  will be calculated from 1-week continuous glucose monitoring data
percent time spent below the glycemic target of 70 mg/dl | week 0 and 12
  will be calculated from 1-week continuous glucose monitoring data
percent time in hypoglycemia below 54 mg/dl | week 0 and 12
  will be calculated from 1-week continuous glucose monitoring data
percent time spent above the glycemic target of 140 mg/dl | week 0 and 12
  will be calculated from 1-week continuous glucose monitoring data
percent time spent in hyperglycemia | week 0 and 12
  will be calculated from 1-week continuous glucose monitoring data
blood glucose average | week 0 and 12
  will be calculated from 1-week continuous glucose monitoring data
blood glucose standard deviation | week 0 and 12
  will be calculated from 1-week continuous glucose monitoring data
Glycemic Variability Index, a measure for glycemic variability normalized to mean blood glucose level | week 0 and 12
  will be calculated by dividing blood glucose standard deviation by blood glucose average
Mean Amplitude of Glycemic Excursions (MAGE), a measure for postprandial glycemic variability | week 0 and 12
  will be calculated by dividing blood glucose standard deviation by blood glucose average
fasting total cholesterol | week 0 and 12
  from venous blood
fasting high density lipoprotein cholesterol | week 0 and 12
  from venous blood
fasting low density lipoprotein cholesterol | week 0 and 12
  from venous blood
fasting triglycerides | week 0 and 12
  from venous blood
fasting beta hydroxybutyrate | weeks 0, 1, 2, 4, 6, 9, 12
  from venous blood and/or point-of-care testing
fasting high-sensitivity c-reactive protein | week 0 and 12
  from venous blood
Self-reported quality of life assessed per self-report by The Problem Areas in Diabetes Scale (PAID) | week 0, 6, and 12
  The scores for each item are summed, then multiplied by 1.25 to generate a total score out of 100.
Becks Depression Inventory II (BDI II) less suicidality | week 0, 6, and 12
  BDI-II less suicidality is a 20-item self-report inventory that measures assesses for presence and severity of depression depressive symptoms. Each item is scored between 0-3. Item scores are added up to a total score (max. 60) and reported.
Yale Food Addiction Scale 2.0 (YFAS 2.0) | week 0, 6, and 12
  Assesses indicators of addictive-like eating.The YFAS includes two scoring options: 1) a "symptom count" that reflects the number of addiction-like criteria endorsed and 2) a dichotomous "diagnosis" that indicates whether a threshold of three or more "symptoms" plus clinically significant impairment or distress has been met. The diagnosis score will be calculated at baseline and used as an effect modifier. Symptom counts will be reported separately as a longitudinal measure.
Highly Processed Food Withdrawal Scale (ProWS) | Baseline, daily on days 1-7, then weekly; primary focus on change from baseline to day 7
  Assesses withdrawal-type symptoms that may occur when individuals cut down on rewarding foods.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lennerz BS, Barton A, Bernstein RK, Dikeman RD, Diulus C, Hallberg S, Rhodes ET, Ebbeling CB, Westman EC, Yancy WS Jr, Ludwig DS. Management of Type 1 Diabetes With a Very Low-Carbohydrate Diet. Pediatrics. 2018 Jun;141(6):e20173349. doi: 10.1542/peds.2017-3349. Epub 2018 May 7. PMID 29735574